CLINICAL TRIAL: NCT04411992
Title: The Effect of Vibration Stimulation on Intramuscular Injection Pain and Patient Satisfaction: A Single-Blind, Randomized Cross-over Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Berna Dincer, Assistant Prof., Istanbul Medeniyet University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 42432570
Record Dates: First submitted 2020-05-29; First posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-06

CONDITIONS: Pain
Keywords: Vibration; Pain management; satisfaction
MeSH Terms: conditions — Pain; Agnosia; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: Two groups were formed according to crossover design. The groups of the patients were determined according to the randomization list formed by using the following website; www.randomization.com.All the measurement scores were obtained by another researcher blinded to group allocation.
Who Masked: Investigator
Masking Description: All the measurement scores were obtained by another researcher blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Allocated to Vibration intervention (1) A (Experimental): Patient information form, visual pain form and satisfaction scale were applied before injection application for all of the patients. The height, weight and BMI of the patients will be measured by the attending nurse. Intramuscular antibiotic injection with vibration will be applied to the ventrogluteal region of the patients .
  Interventions: Device: Vibrating Device
- Allocated to Control intervention (1) B (No Intervention): The height, weight and BMI of the patients will be measured by the attending nurse. Intramuscular antibiotic injection without vibration will be applied to the ventrogluteal region of the patients.
- Allocated to Vibration intervention (2) B (Experimental): Patient information form, visual pain form and satisfaction scale were applied before injection application for all of the patients. The height, weight and BMI of the patients will be measured by the attending nurse. Intramuscular antibiotic injection with vibration will be applied to the ventrogluteal region of the patients .
  Interventions: Device: Vibrating Device
- Allocated to Control intervention (1) A (No Intervention): The height, weight and BMI of the patients will be measured by the attending nurse. Intramuscular antibiotic injection without vibration will be applied to the ventrogluteal region of the patients.

INTERVENTIONS:
Device: Vibrating Device — The device used for the vibration application was produced to control pain and distract attention by providing vibration of 150 at 183 Hz (9000-11,000/min). The device is used again by being cleaned with 70% alcohol. The device was placed put 3 cm above the injection site. It should be ensured to completely contact with skin. Vibration was applied on the site for 3 minutes before injection
  Arms: Allocated to Vibration intervention (1) A; Allocated to Vibration intervention (2) B

SUMMARY:
Intramuscular (IM) injection is the most frequently used nursing practice in the clinic.1 16 billion treatments are performed through injection per year all over the world. Approximately 95% of these injections are administered for therapeutic purpose. There is no study result in the literature on the effect of vibration on pain in the ventrogluteal region in particular.

DETAILED DESCRIPTION:
Intramuscular (IM) injection is the most frequently used nursing practice in the clinic.1 16 billion treatments are performed through injection per year all over the world. Approximately 95% of these injections are administered for therapeutic purpose.

If IM injections are not administered properly, they cause many complications such as primarily pain and cellulitis, muscular fibrosis and contracture, abscesses, tissue necrosis, granuloma, hematoma, and nerve injuries.Painful injections may lead to the development of fear and needle phobia. People are not able to comply with the treatment due to fear and needle phobia and they may even reject treatment. Pain developing after IM injection may vary based on drug content, individual factors and injection technique.

It has been reported that patients feel less pain and the other complications decrease when the correct technique of IM injection is selected. Different pain relief methods such as local ice application, changing needle before injection and acupressure are employed during injection. In the literature, mechano-analgesia, which is known as the skin stimulation methods, is included in pain management in addition to these methods.

One of the mechano-analgesia methods is vibration. The pain-relief mechanism of vibration is explained with the gate control theory. The theory, which is a similar mechanism used to obtain pain relief by rubbing an area near an injury, using TENS, or acupuncture. In the studies, it has been explained by the fact that the sense of touch and vibration obtained from skin receptors stimulate the intermediary inhibitor neurons in medulla spinalis through A-β nerve fibres. These neurons reduce the pain level in A-delta and A-C fibres in transmitting the signal received from skin to the second neuron, the signal cross over medulla spinalis and rises to brain. There are studies in the literature explaining that pain is reduced by vibration. Also, the vibration has advantages over other methods such as TENS, acupuncture as it is a method that is easy to apply, simple, applicable in all hours, and cheap and does not require any preparation.

Although the results of the related studies have indicated that this new method is effective in reducing injection pain, the number of studies on this method in the literature is limited. There is no study result in the literature on the effect of vibration on pain in the ventrogluteal region in particular.

Purpose of the study The purpose of this study was to assess the effect of vibration stimulation application in ventrogluteal region on intramuscular injection pain and patient satisfaction.

The specific study questions were as follows:

1. What are the effects of vibration on intramuscular injection-induced pain?
2. What are the effects of vibration on satisfaction for intramuscular injection?

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and over
* had no communication problem,
* had a body mass index (BMI) of 18.5 to 30 kg/m2,
* not injected in ventrogluteal region in the last two weeks
* not have any pain, hematoma, necrosis, scar, incision or infection symptoms on skin in ventrogluteal region

Exclusion Criteria:

* Have ppain, hematoma, necrosis, scar, incision or infection symptoms on skin in ventrogluteal region
* injected in ventrogluteal region in the last two weeks
* not want to participate.
* body mass index (BMI) of under 18.5 and up 30 kg/m2,
* have psychological illness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2020-06-05 (Estimated); Primary Completion 2020-09-05 (Estimated); Study Completion 2020-09-10 (Estimated)

PRIMARY OUTCOMES:
the effects of vibration on intramuscular injection-induced pain | Three months
  Pain will be measures with Visual Analog Scale (VAS). The scale is composed of a 10-cm vertical or horizontal line, which starts with "No pain" on the one edge and ends with "worst pain" on the other edge. Patients should be informed about the use of VAS very well. Patients are asked to indicate the pain level by marking the appropriate point on the line.
the effects of vibration on satisfaction for intramuscular injection | Three months
  patient satisfaction will be measured with Visual Analog Patient Satisfaction Scale .Visual patient satisfaction scale is combined with the characteristics of the well-known VAS (Visual Analog Scale). It is composed of a 100-mm horizontal line without numbers.

IPD SHARING:
Plan to Share IPD: No